CLINICAL TRIAL: NCT06965842
Title: The Video System to Provide a Developmental Training Guide for In-home, Parent-centered, Early Intervention in Preterm Infants: A Proof of Concept and Feasibility Study
Brief Title: The Video System to Provide a Developmental Training Guide for Preterm Infants
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Woo Hyung Lee, Clinical Associate Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0420222050
Record Dates: First submitted 2025-04-21; First posted 2025-05-11 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Premature Infants; Very Low Birth Weight Infants
Keywords: developmental training; premature infants; very low birth weight infants; early intervention
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention (Experimental)
  Interventions: Other: Parent-centered developmental training

INTERVENTIONS:
Other: Parent-centered developmental training — After discharge from the neonatal intensive care unit, 1:1 monitoring is conducted at home for 30 minutes twice a week using a video conferencing platform (Zoom) until the corrected age of 6 months to provide parent-centered early intervention. Parents film the developmental training process using a smartphone and send the video to the therapist, who analyzes the video data to provide new treatment goals and guidelines.

SUMMARY:
This study aimed to establish a systematic developmental training guide protocol for parent-centered early intervention and verify the concept and feasibility of a video system for parent-centered in-home developmental therapy under the monitoring of a therapist. The target group is premature infants under 32 weeks of gestation or very low birth weight infants under 1500 g with brain damage. A single-arm intervention group of 10 people was recruited, and considering a dropout rate of 20%, the total number of participants was calculated to be 12. 1:1 monitoring to provide parent-centered early intervention at home after discharge from the neonatal intensive care unit is conducted twice a week for 30 minutes per session using a video platform (Zoom) until the corrected age of 6 months. Parents record the developmental training process using a smartphone and transmit it to the therapist, who analyzes the video data to provide new treatment goals and guidelines. Feasibility assessment included: 1) Exercise diary: Number of total and average sessions performed (N) and percentage (%), number of total and average sessions completed (N) and percentage (%) 2) Parent questionnaire 3) Video analysis: Periodic video education and developmental training video acquisition and analysis 4) Heart rate analysis: Analysis of average heart rate during and after rest and developmental training 5) Safety analysis: Number of times (N) and reasons for exercise interruption during developmental training 6) Developmental assessment: Implementation of developmental assessments such as GMOS, MOS-R, HINE, GMFM, and BSID. For safety assessment, if the following symptoms appear during development training, stop exercising and rest until stable. If oxygen saturation drops by more than 10% compared to resting, causing cyanosis and dyspnea, or if heart rate increases by more than 150 beats/min.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants less than 32 weeks of gestation or extremely low birth weight infants less than 1500 g
* Premature infants with a corrected age of less than 1 month
* Brain damage through brain imaging (e.g. cranial USG, brain MRI)

Exclusion Criteria:

* Multiple malformations or genetic abnormalities
* Severe visual or hearing impairment
* Loss of consciousness
* Tracheostomy
* Medically unstable condition

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Number of total and average sessions performed (N) | up to corrected age 6 months
Percentage of total and average sessions performed (%) | up to corrected age 6 months
Number of total and average sessions completed (N) | up to corrected age 6 months
Percentage of total and average sessions completed (%) | up to corrected age 6 months
Parent questionnaire | at corrected age 6 months
General Movement Optimality Score | corrected age 0, 1.5months
  Minimum score: 5 Maximum score: 42 Assessing the quality of writhing movements in infants (typically from term age to 6-9 weeks post-term). Higher scores reflect more optimal general movements - smooth, variable, and age-appropriate. Lower scores may suggest abnormal or poor-quality movements, which are associated with neurological risk.
Motor Optimality Score-Revised | corrected age 4months
  Minimum score: 5 Maximum score: 28
  Evaluating fidgety movements and other spontaneous motor patterns in infants (typically from 9 to 20 weeks post-term). Higher scores indicate better motor repertoire and neurological function, and are associated with typical development. Lower scores are often seen in infants at risk for motor disorders, such as cerebral palsy.
Hammersmith Infant Neurological Examination | corrected age 4, 6, 9 months
  Total Score Range:
  Minimum: 0 Maximum: 78
  The total score is the sum of scores across 26 items, each scored from 0 to 3:
  0 = severely abnormal
  1. = moderately abnormal
  2. = mildly abnormal
  3. = normal Higher HINE scores (closer to 78) indicate better neurological function. Lower scores may suggest neurological impairment or risk for conditions such as cerebral palsy.
Gross Motor Function Measure | corrected age 6, 9 months
  GMFM-88
  Items: 88 items across 5 dimensions:
  Lying and Rolling Sitting Crawling and Kneeling Standing Walking, Running, and Jumping Scoring per item: 0 to 3
  Total Score Range:
  Minimum: 0% Maximum: 100% (Expressed as a percentage of the maximum possible score) Higher scores represent better gross motor function.
Bayley Scales of Infant and Toddler Development | corrected age 9 months
  1. Scaled Scores (for subtests like Fine Motor, Expressive Language, etc.):
     Range:
     Minimum: 1 Maximum: 19 Mean: 10 Standard Deviation (SD): 3
  2. Composite Scores (for broader domains like Cognitive, Motor, etc.):
  Range:
  Minimum: 40 Maximum: 160 Mean: 100 Standard Deviation (SD): 15 130 and above Very Superior 120-129 Superior 110-119 High Average 90-109 Average 80-89 Low Average 70-79 Borderline Below 70 Extremely Low / Delayed
Number of exercise interruption (N) | up to corrected age 6 months
Number of adverse event (N) | up to corrected age 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: No